CLINICAL TRIAL: NCT00310843
Title: A Case-Control Toxicogenomics Study to Identify Unique Genetic Polymorphisms in Patients Who Have Experienced Symptomatic Hepatotoxicity or Severe Cutaneous Toxicity Within the First 8 Weeks of Nevirapine Therapy
Brief Title: Case-Control Viramune (Nevirapine) Toxicogenomics Study
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Other Study IDs: 1100.1452; 2005-004321-26
Record Dates: First submitted 2006-03-28; First posted 2006-04-05 (Estimated); Last update posted 2013-08-01 (Estimated); Status verified 2013-07

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Nevirapine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- All study population
  Interventions: Drug: Nevirapine

INTERVENTIONS:
Drug: Nevirapine — Patients with HIV-1 infection who have taken or are currently taking nevirapine

SUMMARY:
Attempt to identify genetic polymorphisms in interrogated pathways which may be associated with symptomatic hepatotoxicity or severe cutaneous toxicity observed in case patients within the first 8 weeks of nevirapine therapy.

ELIGIBILITY:
Inclusion Criteria:

Inclusion for Case

1. Male or female patients >=18 years of age with HIV-1 infection who experienced one or more of the following adverse reactions within the first 8 weeks of starting nevirapine therapy:

   * Grade 3 or 4 LFT elevation (ALT or AST > 5X ULN) and any symptom consistent with clinical hepatitis (see Appendix 10.1)
   * Acute liver failure secondary to nevirapine therapy*
   * Functional group III or IV rash
   * *Acute liver failure is defined as serious liver injury usually requiring hospitalization that may lead to death or liver transplantation.

   Inclusion for Control
2. Male or female patients >=18 years of age with HIV-1 infection who have been exposed to nevirapine therapy for at least 18 weeks and who do not meet any of the case inclusion criteria

Exclusion Criteria:

Exclusion for Cases

1. Patients with any hepatotoxicity or rash event which in the investigators judgement is not related to nevirapine use (ex. hepatotoxicity due to alcohol or other medicinal use or rash due to other medicinal use).
2. Patients who began abacavir or TMP-SMX (trimethoprim/sulfamethoxazole) therapy 2 weeks or less prior to or up to 8 weeks after initiating nevirapine therapy.
3. Patients with AST or ALT elevations > 5 times the ULN (>= Grade 3) just prior to the initiation of nevirapine therapy.

   Exclusion for Controls
4. Patients who discontinued nevirapine before completing 18 weeks of dosing with 200 mg/day for 2 weeks followed by 400 mg/day thereafter.
5. Patients who developed functional group I, IIa or IIb rash within 18 weeks of starting nevirapine therapy, or any dermatologic condition that could plausibly be attributed to nevirapine.
6. Patients with ALT or AST elevations >2.5 X ULN (>Grade 1) within 18 weeks of starting nevirapine therapy.
7. Any hepatobiliary adverse event that could possibly be attributed to nevirapine.
8. Patients who develop any systemic reaction attributable to nevirapine use during the first 18 weeks of nevirapine treatment such as flu-like symptoms, arthralgia, myalgia, or conjunctivitis.

   Exclusion for Cases and Controls
9. Patients who have participated in the 2NN-Long-term Follow-up study (1100.1454)
10. Patients with CD4 count 150 cells/mm3 prior to the initiation of nevirapine therapy (last available result measured 6 months prior to the initiation of nevirapine therapy).
11. Evidence of acute co-infection with viral hepatitis.
12. Patients taking prednisone, prednisolone, or immuno-modulatory medication within the first 8 weeks of nevirapine therapy.
13. Patients who are unwilling to provide blood samples for DNA testing.
14. Patients who did not sign informed consent and or authorization to release protected health information per local requirements.
15. Patients without available liv

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients Who Have Experienced Symptomatic Hepatotoxicity or Severe Cutaneous Toxicity Within the First 8 Weeks of Nevirapine Therapy
Sampling Method: Non-Probability Sample
Enrollment: 889 (Actual)
Dates: Start 2006-02; Primary Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Endpoints: relationship between nevirapine-related AEs and genetic polymorphisms loci: Drug metabolizing enzymes (e.g., cytochrome P450 isoforms) Drug transporters (e.g., MDR1 and OATP-C) Human Major Histocompatibility Complex region genes

SECONDARY OUTCOMES:
Descriptive demographics comparing cases with matched controls in an attempt to link genetic polymorphisms associated with symptomatic hepatotoxicity or severe cutaneous toxicity (cases) to gender, race or other patient characteristics.

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (102):
- United States (12):
  - 1100.1452.01006 Boehringer Ingelheim Investigational Site, Birmingham, Alabama
  - 1100.1452.01013 Boehringer Ingelheim Investigational Site, Denver, Colorado
  - 1100.1452.99999 Boehringer Ingelheim Investigational Site, Baltimore, Connecticut
  - 1100.1452.01011 Boehringer Ingelheim Investigational Site, New Haven, Connecticut
  - 1100.1452.01003 Boehringer Ingelheim Investigational Site, Baltimore, Maryland
  - 1100.1452.01002 Boehringer Ingelheim Investigational Site, Boston, Massachusetts
  - 1100.1452.01014 Boehringer Ingelheim Investigational Site, Springfield, Massachusetts
  - 1100.1452.01015 Boehringer Ingelheim Investigational Site, St Louis, Missouri
  - 1100.1452.01016 Boehringer Ingelheim Investigational Site, New York, New York
  - 1100.1452.01012 Boehringer Ingelheim Investigational Site, Chapel Hill, North Carolina
  - 1100.1452.01001 Boehringer Ingelheim Investigational Site, Nashville, Tennessee
  - 1100.1452.01004 Boehringer Ingelheim Investigational Site, Fort Worth, Texas
- Argentina (4):
  - 1100.1452.54001 Fundación Huésped, Capital Federal
  - 1100.1452.54002 Funcei, Capital Federal
  - 1100.1452.54003 Boehringer Ingelheim Investigational Site, Capital Federal
  - 1100.1452.54004 Boehringer Ingelheim Investigational Site, Rosario
- Australia (7):
  - 1100.1452.61004 Boehringer Ingelheim Investigational Site, Darlinghurst, New South Wales
  - 1100.1452.61005 Boehringer Ingelheim Investigational Site, Darlinghurst, New South Wales
  - 1100.1452.61006 Boehringer Ingelheim Investigational Site, Darlinghurst, New South Wales
  - 1100.1452.61003 Boehringer Ingelheim Investigational Site, Miami, Queensland
  - 1100.1452.61002 Boehringer Ingelheim Investigational Site, Carlton, Victoria
  - 1100.1452.61008 Boehringer Ingelheim Investigational Site, Melbourne, Victoria
  - 1100.1452.61001 Boehringer Ingelheim Investigational Site, South Yarra, Victoria
- Canada (3):
  - 1100.1452.01501 St. Paul's Hospital, Vancouver, British Columbia
  - 1100.1452.01504 Boehringer Ingelheim Investigational Site, Vancouver, British Columbia
  - 1100.1452.01502 Toronto General Hospital, Toronto, Ontario
- France (33):
  - 1100.1452.3304A Hôpital Saint André, Bordeaux
  - 1100.1452.3306A Hôpital Hôtel Dieu, Lyon
  - 1100.1452.3306B Hop Hôtel Dieu, Lyon
  - 1100.1452.3311A Hôpital Edouard Herriot, Lyon
  - 1100.1452.3311B Pavillon P, Lyon
  - 1100.1452.3311C Hôpital Edouard Herriot, Lyon
  - 1100.1452.3311D Hôpital Edouard Herriot, Lyon
  - 1100.1452.3305A Hôpital hôtel Dieu, Nantes
  - 1100.1452.3305B Hôpital hôtel Dieu, Nantes
  - 1100.1452.3305C Hôpital hôtel Dieu, Nantes
  - 1100.1452.3305D Hôpital Hôtel Dieu, Nantes
  - 1100.1452.3305E Hôpital hôtel Dieu, Nantes
  - 1100.1452.3305F Hôpital Hôtel Dieu, Nantes
  - 1100.1452.3305G Hôpital Hôtel Dieu, Nantes
  - 1100.1452.3305H Hôpital hôtel Dieu, Nantes
  - 1100.1452.3305I Hôpital Hôtel Dieu, Nantes
  - 1100.1452.3301A Hôpital Saint Louis, Paris
  - 1100.1452.3302A Hôpital Tenon, Paris
  - 1100.1452.3303A Hôpital de la Pité Salpêtrière, Paris
  - 1100.1452.3310A Hôpital Bichat Claude Bernard, Paris
  - 1100.1452.3310B Hôpital Bichat Claude Bernard, Paris
  - 1100.1452.3313A Hôpital Saint Antoine, Paris
  - 1100.1452.3313B Hôpital Saint Antoine, Paris
  - 1100.1452.3313C Hôpital Saint Antoine, Paris
  - 1100.1452.3314A Hôpital Européen Georges Pompidou, Paris
  - 1100.1452.3308A Hôpital Purpan, Toulouse
  - 1100.1452.3308B Hôpital Purpan, Toulouse
  - 1100.1452.3307A Hôpital Guy Chateliez, Tourcoing
  - 1100.1452.3307B Hôpital Guy Chateliez, Tourcoing
  - 1100.1452.3307C Hôpital Guy Chateliez, Tourcoing
  - 1100.1452.3307D Hôpital Guy Chateliez, Tourcoing
  - 1100.1452.3307E Hôpital Guy Chateliez, Tourcoing
  - 1100.1452.3312A Hôpital Brabois, Vandœuvre-lès-Nancy
- Germany (13):
  - 1100.1452.4901 Boehringer Ingelheim Investigational Site, Berlin
  - 1100.1452.4902 Boehringer Ingelheim Investigational Site, Berlin
  - 1100.1452.9907 Boehringer Ingelheim Investigational Site, Berlin
  - 1100.1452.4903 Boehringer Ingelheim Investigational Site, Bochum
  - 1100.1452.4918 Boehringer Ingelheim Investigational Site, Bonn
  - 1100.1452.4912 Boehringer Ingelheim Investigational Site, Düsseldorf
  - 1100.1452.4904 Boehringer Ingelheim Investigational Site, Essen
  - 1100.1452.4933 Boehringer Ingelheim Investigational Site, Frankfurt am Main
  - 1100.1452.4916 Boehringer Ingelheim Investigational Site, Hamburg
  - 1100.1452.4931 Boehringer Ingelheim Investigational Site, Hamburg
  - 1100.1452.4910 Boehringer Ingelheim Investigational Site, München
  - 1100.1452.4900 Universitätsklinikum Ulm, Ulm
  - 1100.1452.4932 Boehringer Ingelheim Investigational Site, Würzburg
- Netherlands (2):
  - 1100.1452.31001 Academisch Medisch Centrum, Amsterdam
  - 1100.1452.31002 Onze Lieve Vrouwen Gasthuis, Amsterdam
- Spain (10):
  - 1100.1452.34005 Boehringer Ingelheim Investigational Site, Badalona
  - 1100.1452.34001 Boehringer Ingelheim Investigational Site, Barcelona
  - 1100.1452.34002 Boehringer Ingelheim Investigational Site, Barcelona
  - 1100.1452.34004 Boehringer Ingelheim Investigational Site, Barcelona
  - 1100.1452.34003 Boehringer Ingelheim Investigational Site, L'Hospitalet de Llobregat
  - 1100.1452.34006 Boehringer Ingelheim Investigational Site, Madrid
  - 1100.1452.34007 Boehringer Ingelheim Investigational Site, Madrid
  - 1100.1452.34010 Boehringer Ingelheim Investigational Site, Madrid
  - 1100.1452.34011 Boehringer Ingelheim Investigational Site, Madrid
  - 1100.1452.34009 Boehringer Ingelheim Investigational Site, Seville
- Taiwan (6):
  - 1100.1452.88602 Kaohsiung Veterans General Hospital, Kaohsiung City
  - 1100.1452.88603 E-Da Hospital, Kaohsiung City
  - 1100.1452.88605 Chung-Ho Memorial Hospital, Kaohsiung Medical University, Kaohsiung City
  - 1100.1452.88606 China Medical University Hospital, Taichung
  - 1100.1452.88601 National Taiwan University Hospital, Taipei
  - 1100.1452.88604 Taipei City Hospital, Taipei
- Thailand (3):
  - 1100.1452.66001 Boehringer Ingelheim Investigational Site, Bangkok
  - 1100.1452.66002 Boehringer Ingelheim Investigational Site, Bangkok
  - 1100.1452.66003 Boehringer Ingelheim Investigational Site, Khon Kaen
- United Kingdom (9):
  - 1100.1452.44006 Boehringer Ingelheim Investigational Site, Birmingham
  - 1100.1452.44004 Boehringer Ingelheim Investigational Site, Brighton
  - 1100.1452.44001 Boehringer Ingelheim Investigational Site, Coventry
  - 1100.1452.44002 Boehringer Ingelheim Investigational Site, London
  - 1100.1452.44005 Boehringer Ingelheim Investigational Site, London
  - 1100.1452.44008 Boehringer Ingelheim Investigational Site, London
  - 1100.1452.44009 Boehringer Ingelheim Investigational Site, London
  - 1100.1452.44003 Boehringer Ingelheim Investigational Site, Manchester
  - 1100.1452.44007 Boehringer Ingelheim Investigational Site, Plaistow, London